CLINICAL TRIAL: NCT06539156
Title: Pattern of Prescribing Anticoagulants As DVT Prophylaxis in Intensive Care Unit of Tertiary Hospital
Brief Title: Prescribing Appropriateness of Thrombo-prophylaxis in Intensive Care Unit of Tertiary Hospital
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Egyptian Chinese University (Other); Teachers Hospital (Unknown)
Responsible Party: Principal Investigator, Sarah Sabry Hashem, Clinical Pharmacy Associate Professor, Egyptian Chinese University
Other Study IDs: 2887764466
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: DVT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Medical Patients
  Interventions: Other: DVT prophyllaxis
- Surgical Patients
  Interventions: Other: DVT prophyllaxis

INTERVENTIONS:
Other: DVT prophyllaxis — VTE prophylaxis administration among patients based on the American College of Chest Physicians (ACCP) recommendations

SUMMARY:
Hospitalized patients are at high risk of venous thromboembolism (VTE), and the appropriate use of thromboprophylaxis can significantly reduce the incidence of VTE in high-risk patients. We investigated the pattern of VTE prophylaxis administration among elderly medical patients and assessed its appropriateness based on the American College of Chest Physicians (ACCP) recommendations. Methods A cross-sectional single-center study will be conducted between July 2024 and December 2024, including hospitalized (> 48 h), (≥ 60 years), medical and surgical patients, and excluding patients receiving anticoagulant for other reason, having contraindication to thromboprophylaxis, or had VTE diagnosed within 48 h. The Padua and caprine prediction scores will be used to determine the patients' risk for VTE, and thromboprophylaxis use will be assessed against the ACCP recommendations.

ELIGIBILITY:
Inclusion Criteria:

Patient records

* admitted to the ICU with
* medical or surgical causes
* recieved anticoagulants for DVT prophylaxis

Exclusion Criteria:

* Patients already on anticoagulant therapy,
* had history of previous DVT,
* had End-stage liver disease,
* admitted with hemorrhage/bleeding
* not prescribed DVT prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient records admitted to the ICU with medical or surgical causes treated with anticoagulants for DVT prophylaxis will be collected Patients already on anticoagulant therapy, had history of previous DVT, had End-stage liver disease, admitted with hemorrhage/bleeding or not prescribed DVT prophylaxis will be excluded.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Padua score for medical patients | within 24 hours of ICU admission
  Venous thromboembolism Risk assessment (Scores 0-3 are low risk and do not warrant prophylaxis. Scores ≥4 are high risk for VTE and subsequent complications; recommendation for thromboprophylaxis.)
Caprini score for surgical patients | within 24 hours of ICU admission
  Venous thromboembolism Risk assessment (Total score of 0-1: Low risk of VTE Total score of ≥3: High/moderate risk of VTE )

SECONDARY OUTCOMES:
Bleeding risk assessment | within 24 hours of ICU admission
Direct Anticoagulant cost | within 24 hours of ICU admission till ICU discharge(at least 48 hours)
  sum of costs related to the anticoagulant administration for DVT Prophylaxis
Adverse drug reaction cost | within 24 hours of ICU admission till ICU discharge (at least 48 hours)
  sum of costs related to the Adverse drug reaction for DVT Prophylaxis

CONTACTS AND LOCATIONS:
Locations (1):
- Teachers Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No